CLINICAL TRIAL: NCT05389696
Title: Clinical Trial to Evaluate Safety, Tolerability and Pharmacokinetic Characteristics of MIT-001 After Subcutaneous and Intravenous Administration in Healthy Subjects
Brief Title: Clinical Trial to Evaluate Pharmacokinetic Characteristics of MIT-001 After SC Administration in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MitoImmune Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MIT001-FD-SC01
Record Dates: First submitted 2022-05-10; First posted 2022-05-25 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Heathly Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part1. Group1. MIT-001 SC 10mg (Experimental): Single subcutaneous administration of 10mg MIT-001 or placebo
  Interventions: Drug: Single subcutaneous administration and Blood collection
- Part1. Group2. MIT-001 SC 20mg (Experimental): Single subcutaneous administration of 20mg MIT-001 or placebo
  Interventions: Drug: Single subcutaneous administration and Blood collection
- Part1. Group3. MIT-001 SC 40mg and IV 40mg (Experimental): Single subcutaneous administration of 40mg MIT-001 or placebo and then signle intravenous administration of 40mg MIT-001 or placebo
  Interventions: Drug: Single subcutaneous administration and then IV injection.
- Part2. Group1: MIT-001 SC 20mg (Experimental): Multiple subcutaneous administration of 20mg MIT-001/day or placebo for 7days
  Interventions: Drug: MIT-001 20mg and 40mg_Multiple administration
- Part2. Group2: MIT-001 SC 40mg (Experimental): Multiple subcutaneous administration of 40mg MIT-001/day or placebo for 7days
  Interventions: Drug: MIT-001 20mg and 40mg_Multiple administration

INTERVENTIONS:
Drug: Single subcutaneous administration and Blood collection — Single subcutaneous administration and Blood collection
  Other Names: MIT-001 10mg and 20mg
  Arms: Part1. Group1. MIT-001 SC 10mg; Part1. Group2. MIT-001 SC 20mg
Drug: Single subcutaneous administration and then IV injection. — Single subcutaneous administration and then single intravenous administration after 2 weeks. In addition Blood collection is conducted as scheduled.
  Other Names: MIT-001 40mg
  Arms: Part1. Group3. MIT-001 SC 40mg and IV 40mg
Drug: MIT-001 20mg and 40mg_Multiple administration — Multiple subcutaneous administration for 7 days and then blood collection
  Other Names: MIT-001 20mg and 40mg
  Arms: Part2. Group1: MIT-001 SC 20mg; Part2. Group2: MIT-001 SC 40mg

SUMMARY:
1. Part 1 Randimization, Double blinded, Placebo controlled, Dose escalation(10mg, 20mg, 40mg) of MIT-001 SC or IV single administration to evaluate safety, tolerability and PK in healthy adult.
2. Part2 Randimization, Double blinded, Placebo controlled, MIT-001 SC multiple administration for 7days (20mg & 40mg) to evaluate safety, tolerability and PK in healthy adult.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, single and multiple dose, dose escalation clinical trial in 40 healthy subjects. This study consists of part 1(single dose for group 1, 2, 3) and part 2(multiple dose for 7 days to group 1 and 2). Subjects will be assigned in 6:2 allocation to receive active or placebo treatments. The purpose of this clinical trial is to evaluate the safety, tolerability and pharmacokinetic properties of MIT-001 after single and multiple subcutaneous administration in healthy adults and to compare IV administration.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy adult between 19 and 45 at the time of screening
2. A person who weigh 55.0 kg or more and 90.0 kg or less at the time of screening and have a body mass index (BMI) of 18.0 or more and 27.0 or less

   ☞ BMI (kg/m2) = Weight (kg) / {Height (m)}2
3. A person who voluntarily decides to participate after hearing and fully understanding the detailed explanation of this clinical trial and consents in writing before the screening procedure
4. A person suitable as a test subject for this study when judged by the investigator through physical examination, clinical laboratory examination, questionnaire, etc.

Exclusion Criteria:

1. Clinically significant liver, kidney, nervous system, immune system, respiratory system, endocrine system disease, blood/tumor disease, cardiovascular disease, mental disease (mood disorder, obsessive-compulsive disorder, etc.) or a history of above diseases
2. A person with a history of hypersensitivity or clinically significant hypersensitivity to clinical investigational drugs, drugs containing the same class of ingredients, and other drugs (aspirin, antibiotics, etc.)
3. At screening, QTc > 450 ms on ECG or other clinically significant findings
4. A person with AST and ALT exceeding 1.5 times the upper limit of the normal range during screening
5. A person with eGFR of less than 60 mL/min/1.73m2 measured using the CKD EPI formula in clinical laboratory tests at screening
6. At screening, systolic blood pressure > 160 mmHg or < 90 mmHg, or diastolic blood pressure > 100 mmHg or < 50 mmHg
7. A person with a history of drug abuse or who have tested positive for drugs of abuse in urine drug screening tests
8. A person who has taken any prescription drugs or herbal medicines within 2 weeks before the first scheduled administration date, or have taken any over-the-counter (OTC), health functional food, or vitamin preparations within 1 week In cases where it is reasonable, they can participate in the clinical trial) or those who are expected to take it
9. A person who has taken drugs that induce or inhibit drug metabolizing enzymes, such as barbiturates, within 1 month before the first scheduled administration date
10. A person who has participated in other clinical trials or bioequivalence studies within 6 months prior to the scheduled first administration date and received the investigational drug or bioequivalence study drug
11. A person who has donated whole blood within 2 months before the first scheduled dose or donated component blood within 1 month, or received blood transfusion within 1 month before the first scheduled dose
12. A person who continuously drinks alcohol (more than 21 units/week, 1 unit = 10 g of pure alcohol (≒ 1 glass of soju or 250 mL of beer)) or cannot abstain from alcohol during the clinical trial period
13. Smokers (However, if you quit smoking 3 months before the first scheduled dose, you can be selected as a test subject)
14. A person who has consumed caffeine-containing foods (coffee, tea (black tea, green tea, etc.), carbonated drinks, coffee milk, nourishing drinks, etc.) within 24 hours of hospitalization for clinical trials and those who cannot refrain from consuming them during hospitalization
15. A person who does not use the following medically acceptable contraceptive methods for 1 month from participation in the clinical trial to the last administration of the investigational drug A. Use of an intrauterine device (copper loop, hormone-containing intrauterine system) with a proven rate of pregnancy failure in the spouse (or partner) B. Concomitant use of either a spermicide or a parenteral hormonal contraceptive with a barrier contraceptive method (male or female) C. Surgery of you or your partner (vasectomy, fallopectomy/ligation, hysterectomy, etc.) D. Use of a cervical cap or contraceptive diaphragm with a male condom
16. Pregnant or lactating women
17. A person who judged the investigator to be inappropriate to participate in the clinical trial due to other reasons

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
PK_Cmax_Part1 Group 1&2 | Part1. Group 1&2: Before SC administration(Day0, 0hour) to 144hour after administration 16 points.
  Part 1, Group 1,2: Cmax
PK_Cmax_Part1 Group 3 | Part1. Group 3_Before SC administration(Day0, 0hour) to 144hour 16 points and then Before IV administration on 15th day(0hour) to 144hour after IV administration 17points.
  Part 1, Group 3: Cmax
PK_AUClast_Part1 Group 1&2 | Part1. Group 1&2_Before SC administration(Day0, 0hour) to 144hour after administration 16 points.
  Part1, Group 1&2: AUClast
PK_AUClast_Part1 Group 3 | Part1. Group 3_Before SC administration(Day0, 0hour) to 144hour 16 points and then Before IV administration on 15th day(0hour) to 144hour after IV administration 17points.
  Part 1, Group 3: AUClast
PK_AUCinf_Part 1, Group 1&2 | Part1. Group 1&2_Before SC administration(Day0, 0hour) to 144hour after administration 16 points.
  Part 1, Group 1&2: AUCinf
PK_AUCinf_Part 1, Group 3 | Part1. Group 3_Before SC administration(Day0, 0hour) to 144hour 16 points and then Before IV administration on 15th day(0hour) to 144hour after IV administration 17points.
  Part 1, Group 3: AUCinf
PK_Tmax_Part 1, Group 1&2 | Part1. Group 1&2_Before SC administration(Day0, 0hour) to 144hour after administration 16 points.
  Part 1, Group 1&2: Tmax
PK_Tmax_Part 1, Group 3 | Part1. Group 3_Before SC administration(Day0, 0hour) to 144hour 16 points and then Before IV administration on 15th day(0hour) to 144hour after IV administration 17points.
  Part 1, Group 3: Tmax
PK_t1/2_Part 1, Group 1&2 | Part1. Group 1&2_Before SC administration(Day0, 0hour) to 144hour after administration 16 points.
  Part 1, Group 1&2: t1/2
PK_t1/2_Part 1, Group 3 | Part1. Group 3_Before SC administration(Day0, 0hour) to 144hour 16 points and then Before IV administration on 15th day(0hour) to 144hour after IV administration 17points.
  Part 1, Group 3: t1/2
PK_Vd/F_Part 1, Group 1&2 | Part1. Group 1&2_Before SC administration(Day0, 0hour) to 144hour after administration 16 points.
  Part 1, Group 1&2: Vd/F
PK_Vd/F_Part 1, Group 3 | Part1. Group 3_Before SC administration(Day0, 0hour) to 144hour 16 points and then Before IV administration on 15th day(0hour) to 144hour after IV administration 17points.
  Part 1, Group 3: Vd/F
PK_CL/F_Part 1, Group 1,2 | Part1. Group 1&2_Before SC administration(Day0, 0hour) to 144hour after administration 16 points.
  Part 1, Group 1,2: CL/F
PK_CL/F_Part 1, Group 3 | Part1. Group 3_Before SC administration(Day0, 0hour) to 144hour 16 points and then Before IV administration on 15th day(0hour) to 144hour after IV administration 17points.
  Part 1, Group 3: CL/F
PK_MRT_Part 1, Group 1&2 | Part1. Group 1&2_Before SC administration(Day0, 0hour) to 144hour after administration 16 points.
  Part 1, Group 1,2: MRT
PK_MRT_Part 1, Group 3 | Part1. Group 3_Before SC administration(Day0, 0hour) to 144hour 16 points and then Before IV administration on 15th day(0hour) to 144hour after IV administration 17points.
  Part 1, Group 3: MRT
PK_F_Part1, Group1,2 | Part1. Group 1&2_Before SC administration(Day0, 0hour) to 144hour after administration 16 points.
  Part 1, Group 1,2: F
PK_F_Part1, Group3 | Part1. Group 3_Before SC administration(Day0, 0hour) to 144hour 16 points and then Before IV administration on 15th day(0hour) to 144hour after IV administration 17points.
  Part 1, Group 3: F
PK_Part2_Cmax | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: Cmax
PK_Part2_Cmin | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: Cmin, Cavg, AUCtau, Tmax, t1/2, Vd/F, CL/F, Cmax,ss, Cmin,ss, Cavg,ss, AUCtau,ss, Tmax,ss, t1/2,ss, Vdss/F, CLss/F, PTF, Rac
PK_Part2_Cavg | Par2_Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: Cavg
PK_Part2_AUCtau | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: AUCtau
PK_Part2_Tmax | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: Tmax
PK_Part2_t1/2 | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: t1/2
PK_Part2_Vd/F | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: Vd/F
PK_Part2_CL/F | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: CL/F
PK_Part2_Cmax,ss | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: Cmax,ss
PK_Part2_Cmin,ss | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: Cmin,ss
PK_Part2_Cavg,ss | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: Cavg,ss
PK_Part2_AUCtau,ss | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: AUCtau,ss
PK_Part2_Tmax,ss | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: Tmax,ss
PK_Part2_t1/2,ss | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: _t1/2,ss
PK_Part2_Vdss/F | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: _Vdss/F
PK_Part2_CLss/F | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: _VCLss/F
PK_Part2_PTF | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: _PTF
PK_Part2_Rac | Part2: Before SC administration(Day0, 0hour) to 24hour 13points, Day5 0hour, Day6 0hour and then Day7 0hour to 216hour after SC administration 17points
  Part 2: _Rac

CONTACTS AND LOCATIONS:
Overall Officials: SeungHwan Lee, MD, Principal Investigator — Seoul National University
Locations (1):
- Seoul National University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No